CLINICAL TRIAL: NCT05655260
Title: PErsonalized TReatment for Endometrial Carcinoma
Acronym: PETREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Turku University Hospital (Other Government); Tampere University Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Kymenlaakso Central Hospital Kotka Finland (Other); Päijänne Tavastia Central Hospital (Other); South Carelia Central Hospital (Other)
Responsible Party: Principal Investigator, Mikko Loukovaara, Chief of Specialists, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/2360/2021
Record Dates: First submitted 2022-11-30; First posted 2022-12-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Adenocarcinoma
Keywords: Endometrial carcinoma; Molecular classification; Adjuvant therapy
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Comprehensive cohort design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- p53 abn subtype and nonendometrioid carcinomas (Experimental): p53 abn stage I-II MI (myometrial invasion) >0%; MMR-D/NSMP nonendometrioid stage I-II MI >0%
  Interventions: Other: Comparison of chemotherapy vs. chemoradiotherapy
- MMR-D molecular subgroup (Experimental): MMR-D stage IA-B grade 1-2, substantial LVSI; MMR-D stage IA grade 3, substantial LVSI; MMR-D stage IB grade 3; MMR-D stage II grade 1-3;
  Interventions: Other: Comparison of VBT vs. WPRT
- NSMP molecular subgroup (Experimental): NSMP stage IA-B grade 1-2, substantial LVSI; NSMP stage IA grade 3, substantial LVSI; NSMP stage IB grade 3; NSMP stage II grade 1-3;
  Interventions: Other: Comparison of VBT vs. WPRT

INTERVENTIONS:
Other: Comparison of chemotherapy vs. chemoradiotherapy — Chemotherapy (paclitaxel-carboplatin) vs. chemoradiotherapy (paclitaxel-carboplatin followed by whole pelvic radiotherapy)
  Patients assigned to chemotherapy receive paclitaxel (175 mg/m2) and carboplatin (area under curve, 5) every 3 weeks for 6 cycles. The pelvic radiotherapy dose is 45 to 50.4 Gy over 5 to 6 weeks (1.8 Gy per day for 25 to 28 fractions).
  Arms: p53 abn subtype and nonendometrioid carcinomas
Other: Comparison of VBT vs. WPRT — Vaginal brachytherapy vs. whole pelvic radiotherapy
  Patients randomized to vaginal brachytherapy receive cuff brachytherapy at 21 Gy in 3 fractions of 7 Gy at 0.5 cm depth. The pelvic radiotherapy dose is 45 to 50.4 Gy over 5 to 6 weeks (1.8 Gy per day for 25 to 28 fractions).
  Arms: MMR-D molecular subgroup; NSMP molecular subgroup

SUMMARY:
The goal of this clinical trial is to compare the efficacy of adjuvant therapies in women with stage I-II molecular integrated high-intermediate or high-risk endometrial carcinoma. Specifically, the invesigators want to compare:

* Chemotherapy vs. chemoradiotherapy in p53 abn subtype and nonendometrioid carcinomas.
* Vaginal brachytherapy vs. whole pelvic radiotherapy in the MMR-D molecular subgroup.
* Vaginal brachytherapy vs. whole pelvic radiotherapy in the NSMP molecular subgroup.

DETAILED DESCRIPTION:
Endometrial carcinomas can be classified into four molecular subgroups, i.e. mismatch repair deficient (MMR-D), p53 abnormal (p53 abn), polymerase-ϵ (POLE) ultramutated, and "no specific molecular profile" (NSMP). Molecular subgroups can be considered to be distinct diseases as they are associated with different clinicopathologic characteristics, prognoses and, possibly, responses to adjuvant therapy. Molecular classification of endometrial carcinoma is recommended to be implemented in routine clinical practice to improve prognostication and triage to adjuvant therapy. The PErsonalized TReatment for Endometrial Carcinoma (PETREC) trial, led by the Finnish Gynecologic Oncology Group (FINGOG), is a multicenter prospective clinical trial for women with stage I-II molecular integrated high-intermediate or high-risk endometrial carcinoma. The efficacy of chemotherapy vs. chemoradiotherapy is compared in p53 abn subtype and nonendometrioid carcinomas, and vaginal brachytherapy vs. whole pelvic radiotherapy in MMR-D and NSMP molecular subgroups. Patients who consent to follow-up within the trial but not to randomization are treated as recommended in multidisciplinary meetings and enrolled for follow-up only (comprehensive cohort study design). The primary outcome is the 5-year cumulative incidence of disease recurrence. Secondary outcomes are vaginal, pelvic, and distant recurrence rates, 5-year recurrence-free and overall survival, adverse events, and patient-reported symptoms and quality of life. The findings of the trial may eventually help decrease under- and overtreatment and, consequently, improve patient outcome and decrease treatment-associated adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 100 years
* WHO performance status 0 to 2
* Stage I-II molecular integrated high-intermediate or high-risk endometrial carcinoma

Exclusion Criteria:

* Age <18 years or >100 years
* WHO performance status >2
* Uterine sarcoma
* A history of malignancy within 5 years
* Previous pelvic radiotherapy
* An interval of >30 days between surgery and start of chemotherapy or >8 weeks between surgery and start of radiotherapy (longer intervals may be permitted with investigator´s approval)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility not based on self-representation of gender identity.
Enrollment: 300 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer reappearance | 5 years
  Cumulative incidence of disease recurrence

SECONDARY OUTCOMES:
Location of cancer reappearance | 5 years
  Vaginal, pelvic, and distant recurrence rates
Overall survival | 5 years
  The time from surgery to death
Recurrence-free survival | 5 years
  The time from surgery to cancer recurrence
Adverse events | 5 years
  Adjuvant therapy-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Loukovaara, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loukovaara M, Butzow R, Staff S, Maenpaa M, Faltinova M, Lassus H, Veijalainen O, Gronvall M, Vaalavirta L, Kuikka E, Haataja M, Urpilainen E, Simojoki M, Anttila M, Auranen A. PErsonalized TReatment for Endometrial Carcinoma (PETREC): study design and methods of a prospective Finnish multicenter trial. Int J Gynecol Cancer. 2023 Nov 6;33(11):1807-1811. doi: 10.1136/ijgc-2023-004939. PMID 37813479